CLINICAL TRIAL: NCT04960280
Title: Use of a Computerized Body Auscultation Device (©VoqX) for the Diagnosis of Structural Cardiac Pathologies
Brief Title: A Study to Evaluate a Computerized Stethoscope Called ©Voqx to Diagnose Heart Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rajiv Gulati, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-012844
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Isolated Aortic Stenosis; Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Computerized Auscultation (Experimental): Patients presenting to the echocardiogram laboratory for routine clinically indicated echocardiography or to the cardiac catheterization laboratory for routine clinically indicated catheterization procedures will undergo a computerized auscultation using the ©VoqX stethoscope and will have their heart sounds auscultated and recorded.
  Interventions: Device: ©VoqX stethoscope

INTERVENTIONS:
Device: ©VoqX stethoscope — Computerized auscultation detects both infrasound and audible sounds and is capable of amplifying auscultated sounds by a factor of thirty.

SUMMARY:
The purpose of this study is to determine whether recording heart sounds with an acoustic stethoscope, combined with artificial intelligence (computer information), will show similar abnormalities to an echocardiogram or cardiac catheterization.

DETAILED DESCRIPTION:
In the current study the plan is to recruit 600 patients who have been referred to the echocardiogram laboratory for routine clinically indicated echocardiography, or to the cardiac catheterization laboratory for routine clinically indicated catheterization procedures. Individuals with normal heart structure and sounds, isolated aortic stenosis (of varying severity), and isolated mitral regurgitation (of varying severity) will be included, while excluding individuals who have multiple valve involvements or combined valve pathologies. Each patient will have baseline testing using the ©CompuSteth device, which will be used to auscultate and record each patient's heart sounds at the bedside prior to the index echocardiogram or cardiac catheterization procedure. This process will take less than 10 minutes and is outlined below. Patients will then proceed with their clinically indicated echocardiograms or cardiac catheterization procedures.

Amongst the first 200 study participants, the results of the echocardiograms and invasive cardiac catheterization procedures will be used to train the ©VoqX device to identify normal heart and to screen and grade for various cardiac structural pathologies, aortic stenosis, and mitral regurgitation, diagnosed by gold-standard testing. Subsequently, after the ©VoqX device has been trained how to characterize and identify sounds that correspond to various structural cardiac pathologies, the next step is to prospectively 'test' how well the ©VoqX device is able to screen normal heart from cardiac pathologies, such as aortic stenosis, and mitral regurgitation, and identify the severity of the valve disorder in the subsequent 200 participants of the study. This will be done by comparing the results obtained from auscultation with the ©VoqX device against the results obtained from gold-standard testing with echocardiography or invasive cardiac catheterization.

ELIGIBILITY:
Inclusion Criteria

* Aged 18 years of age or older.
* Referred to the echocardiogram laboratory for routine clinically indicated echocardiography, or to the cardiac catheterization laboratory for routine clinically indicated catheterization procedures
* Individuals with normal heart sounds, isolated aortic stenosis (any degree of severity), or isolated mitral regurgitation (any degree of severity)

Exclusion Criteria

* Patients with unstable cardiovascular or pulmonary disease
* Patients with mixed valvular heart disease, corresponding to more than one type of valve pathology (i.e.: Aortic stenosis and Aortic Regurgitation), or more than 1 valve involved (i.e.: aortic stenosis and mitral regurgitation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
collecting computerized auscultation data in a time-efficient manner at the bedside is feasible | 2 years
  i) As part of the initial part of the study, that collecting computerized auscultation data using the ©CompuSteth device from patients presenting to the echocardiogram laboratory for routine clinically indicated echocardiography, or to the cardiac catheterization laboratory for routine clinically indicated catheterization procedures in a time-efficient manner at the bedside is feasible. Further, that we can successfully train the ©CompuSteth device to screen for normal heart structure and sounds as well as for a variety of structural cardiac pathologies, including aortic stenosis and its severity, and mitral regurgitation and its severity, using echocardiography or invasive cardiac catheterization as gold standard testing for the presence or absence of structural cardiac pathologies

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Gulati, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No